CLINICAL TRIAL: NCT06054321
Title: A Randomized Clinical Trial of Response to Psychopharmacotherapy According to Multimodal Serum Biomarkers in Depressive Patients
Brief Title: Psychopharmacotherapy for Depressive Patients
Acronym: BMDD-2022
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Min Kim, Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BMDD-2022
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder
Keywords: depression; antidepressant monotherapy; stepwise psychopharmacotherapy; multimodal serum biomarker score
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: partial masking(participants, care providers, outcome assessor are not aware of treatment response scores in spite of opened status for prescribed information (mono vs step)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Good responder group-stepwise pharmacotherapy group (Experimental): Using multimodal serum biomarker scores, patients will be divided into good/poor responder. Then good responder group will be randomized into stepwise pharmacotherapy group vs antidepressant monotherapy(escitalopram) group.
  In the stepwise pharmacotherapy group, treatment strategies (augmentation with antipsychotics (aripiprazole), augmentation with mood stabilizer (lithium),combination (mirtazapine)) will be determined every 3 weeks.
  Interventions: Drug: stepwise pharmacotherapy
- Good responder group-antidepressant monotherapy group (Active Comparator): Using multimodal serum biomarker scores, patients will be divided into good/poor responder. Then good responder group will be randomized into stepwise pharmacotherapy group vs antidepressant monotherapy(escitalopram) group.
  In the antidepressant monotherapy group, dosage escalation will be determined every 3 weeks.
  Interventions: Drug: antidepressant monotherapy group
- Poor responder group-stepwise pharmacotherapy group (Experimental): Using multimodal serum biomarker scores, patients will be divided into good/poor responder. Then poor responder group will be randomized into stepwise pharmacotherapy group vs antidepressant monotherapy(escitalopram) group.
  In the stepwise pharmacotherapy group, treatment strategies (augmentation with antipsychotics (aripiprazole), augmentation with mood stabilizer (lithium),combination (mirtazapine)) will be determined every 3 weeks.
  Interventions: Drug: stepwise pharmacotherapy
- Poor responder group-antidepressant monotherapy group (Active Comparator): Using multimodal serum biomarker scores, patients will be divided into good/poor responder. Then poor responder group will be randomized into stepwise pharmacotherapy group vs antidepressant monotherapy(escitalopram) group.
  In the antidepressant monotherapy group, dosage escalation will be determined every 3 weeks.
  Interventions: Drug: antidepressant monotherapy group

INTERVENTIONS:
Drug: stepwise pharmacotherapy — In the stepwise pharmacotherapy group, treatment strategies (augmentation with antipsychotics (aripiprazole), augmentation with mood stabilizer (lithium),combination (mirtazapine)) will be determined every 3 weeks.
  Other Names: escitalopram; escitalopram with aripiprazole augmentation; escitalopram with lithium augmentation; escitalopram with mirtazapine combination
  Arms: Good responder group-stepwise pharmacotherapy group; Poor responder group-stepwise pharmacotherapy group
Drug: antidepressant monotherapy group — In the antidepressant monotherapy group, dosage escalation will be determined every 3 weeks.
  Other Names: escitalopram monotherapy
  Arms: Good responder group-antidepressant monotherapy group; Poor responder group-antidepressant monotherapy group

SUMMARY:
The primary purpose of this study is to compare the short (12 week) and long-term (1-year) efficacy and the tolerability between stepwise psychopharmacotherapy and antidepressant monotherapy for 12 weeks in adult patients with major depressive disorders, stratified by the multimodal serum biomarker scores.

DETAILED DESCRIPTION:
This is prospective randomized controlled trials (RCT) to evaluate clinical impact of antidepressant monotherapy vs stepwise psychopharmacotherapy in patients with major depressive disorders, stratified by multimodal serum biomarker scores. Participants will be predicted treatment response based on the multimodal serum biomarker scores at baseline, will be categorized into good and poor treatment responders and then randomly assigned to two groups: stepwise pharmacotherapy group and antidepressant monotherapy group. The hypothesis is that in the good treatment responder, the depression remission will be achieved irrespective of treatment modality (stepwise pharmacotherapy or antidepressant monotherapy) group while in poor treatment responders, the treatment response of stepwise pharmacotherapy will be superior to those of antidepressant monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 19 to 65 years
* Diagnostic and Statistical Manual of Mental Disorders-IV criteria for major depressive disorder by study psychiatrists
* Score≥17 on Hamilton Depression Rating Scale-17
* With ability to understand the objective of the study and sign informed consent
* Initiation of an antidepressant treatment for the current episode or no psychotropics excluding sleep pills or benzodiazepines within 1 month of participation

Exclusion Criteria:

* Current or lifetime diagnosis of bipolar disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, psychotic disorder not otherwise specified, or other psychotic disorders
* current major depressive disorder with psychotic features
* History of organic psychosis, epilepsy, or seizure disorder
* Current anorexia nervosa or obsessive compulsive disorder
* Unstable or uncontrolled medical condition
* Unable to complete the psychiatric assessment or comply with the medication regimen due to a severe physical illness
* History of anticonvulsant treatment
* Electroconvulsive therapy for the current depressive episode
* Hospitalization for any psychiatric diagnosis except depressive disorder (e.g., alcohol/drug dependence)
* severly high risk of suicide, self-harm or homicide by investigator's assessment
* Pregnant or breastfeeding
* lack of treatment information on the current depressive episode

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Remission and treatment response status by Hamilton Depression Rating Scale | From baseline to 12 week, 1 year
  Remission defined by total scores of Hamilton Depression Rating Scale (0-52; higher score indicates severe symptom) ≤7 and treatment response defined as ≥50% decrease in the baseline total scores of Hamilton Depression Rating Scale after stepwise psychopharmacotherapy or antidepressant monotherapy

SECONDARY OUTCOMES:
The changes of Hamilton Rating Scale for Depression total score | From baseline to 12 week, 1 year
  To measure the change of the severity of depressive symptoms using observer rating scale after stepwise psychopharmacotherapy or antidepressant monotherapy
The changes of Hospital Anxiety and Depression Scale total score, depression subscore, anxiety subscore | From baseline to 12 week, 1 year
  The Hospital Anxiety and Depression Scale will be used to measure the change of the severity of depressive symptoms using observer rating scale after stepwise psychopharmacotherapy or antidepressant monotherapy. This scale consists of 14 items with a total score ranging from 0 to 42 and divided into two subscales: 7 items of the anxiety subscale (HADS-A) and 7 items of the depression subscale (HADS-D). Higher scores indicate more severe symptoms.
The changes of Clinical Global Impression-severity and improvement score | From baseline to 12 week, 1 year
  The Clinical Global Impression-severity and improvement score is used to measure the change of the global severity and improvement of depressive symptoms after stepwise psychopharmacotherapy or antidepressant monotherapy. This scale is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients. Higher scores indicate more severe psychopathology.
The changes of Brief Psychiatric Rating Scale suicide item score | From baseline to 12 week, 1 year
  Suicidality was evaluated with the suicide-related items on the Brief Psychiatric Rating Scale which assesses the level of 18 symptom constructs such as hostility, suspiciousness, hallucination, and grandiosity. Among the 18 items, suicide item that ranges from 1 (not present) to 7 (extremely severe) will be used to measure the change sof suicidality after stepwise psychopharmacotherapy or antidepressant monotherapy.
The changes of EuroQol-5 Dimension score | From baseline to 12 week, 1 year
  To measure the change of quality of life status after stepwise psychopharmacotherapy or antidepressant monotherapy, EuroQol-5 Dimension is used. This scale has five descriptive questions which may have one of three-level answers and a visual analog scale (VAS) on which patients can mark their current health state. visual analog scale (VAS) on which patients can mark their current health state. The 5 Dimension (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) have three levels of functioning each (no problems, some problems, and unable to/extreme problems) while the visual analog scale ranges from 0 (worst imaginable health state) to 100 (best imaginable health state).
The changes of Social and Occupational Functioning Assessment Scale score | From baseline to 12 week
  To measure the change of the social and occupational function after stepwise psychopharmacotherapy or antidepressant monotherapy, Social and Occupational Functioning Assessment Scale is used that ranges from 0 to 100, with lower scores representing lower functioning.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) in the Treatment Period | First dose of study drug to last dose of study drug in the 26-week Treatment Period and 1 year after baseline
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (i.e. laboratory value), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product. A TEAE is an AE that occurs or worsens after receiving study drug

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Min Kim, MD, PhD, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hospital, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: No
Participant data (without individual identification data) will be translated into coded data and will be available from the principal investigator (J-M Kim) upon reasonable request.

REFERENCES:
- [Background] Kim JM, Kang HJ, Kim JW, Jhon M, Choi W, Lee JY, Kim SW, Shin IS, Kim MG, Stewart R. Prospective associations of multimodal serum biomarkers with 12-week and 12-month remission in patients with depressive disorders receiving stepwise psychopharmacotherapy. Brain Behav Immun. 2022 Aug;104:65-73. doi: 10.1016/j.bbi.2022.05.012. Epub 2022 May 23. PMID 35618226